CLINICAL TRIAL: NCT06045819
Title: Study of the Association Between Residual Venetoclax Plasma Concentration and Composite Complete Remission in Adults with Newly Diagnosed Acute Myeloid Leukemia Ineligible for Intensive Chemotherapy (PREDICLAX)
Brief Title: Relation Between Venetoclax Plasma Concentration and Remission in Adults with Acute Myeloid Leukemia (PREDICLAX)
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A01909-36
Record Dates: First submitted 2023-09-04; First posted 2023-09-21 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Blood Specimen Collection; Technology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * plasma is obtained through venipuncture
  * capillary blood is obtained by pricking a finger
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Patients with composite complete remission: Patients in composite complete remission following the first cycle of venetoclax (400 mg/day, orally, after a ramp-up phase of the first 3 days) + azacytidine (75mg/m²,intravenous, at the start of each cycle from day 1 to day 7)
  Interventions: Biological: Blood sampling for venetoclax drug dosage (venous puncture)
- Patients without composite complete remission: Patients not in composite complete remission following the first cycle of venetoclax (400 mg/day, orally, after a ramp-up phase of the first 3 days) + azacytidine (75mg/m²,intravenous, at the start of each cycle from day 1 to day 7)
  Interventions: Biological: Blood sampling for venetoclax drug dosage (venous puncture)

INTERVENTIONS:
Biological: Blood sampling for venetoclax drug dosage (venous puncture) — 8 blood samples for venetoclax and azole antifungal drugs identification and dosage will be taken by venous and capillary punctures throughout management of patients
  Other Names: Biological: Capillary Blood sampling for venetoclax drug dosage with Volumetric Absorptive Microsampling (VAMS™) technology with Mitra® device (CE-IVD /IVDR); Biological: Blood sampling for azole antifungal drug dosage (venous puncture)

SUMMARY:
Background: In combination with hypomethylating drugs, venetoclax has recently changed the therapeutic management of patients with newly diagnosed acute myeloid leukemia (AML) for whom standard induction chemotherapy was not an option. Over and above the clinical benefits of this combination, the data show that more than half the patients did not show remission criteria, even after the first month's exposure to venetoclax.

Hypothesis: To compare the mean residual venetoclax plasma concentrations obtained in patients who went into complete composite remission versus those who did not go into remission at the end of the first cycle of venetoclax + azacitidine treatment.

Method: According to the French law, this is a multicenter, non-comparative, open-label, single-arm, interventional study with minimal risks and constraints. Selection, information and inclusion will concern adult patients (≥60 years) with a confirmed diagnosis of AML according to ELN 2022 guidelines. Included patients will be treated as standard care with a combination of venetoclax+azacitidine. This research protocol will not modify their usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have a confirmed diagnosis of previously untreated AML (ELN 2022 criteria) within 28 days of the onset of symptoms. Only previous cytoreductive treatments (e.g. hydroxyurea) are authorized.
2. Subject must be ineligible for standard cytarabine and anthracycline induction therapy according to the following criteria:

   * Subject aged ≥ 75 years.
   * OR subject aged between 60 and 74 with at least one of the following comorbidities:

     * ECOG performance status: of 2 or 3.
     * cardiac history: heart failure requiring treatment, left ventricular ejection fraction ≤ 50%, chronic stable angina.
     * carbon monoxide diffusion capacity ≤ 65% or forced expiratory volume in one second ≤ 65%.
     * creatinine clearance between 30 and 45 mL/min/m².
     * liver damage (not related to AML) with total bilirubin between 1.5 and 3 × upper normal limit.
     * any other comorbidity deemed by the physician to be incompatible with standard induction chemotherapy.
3. Patients are eligible for the recommended standard treatment, i.e. a combination of venetoclax and a hypomethylating agent.
4. Subjects must voluntarily sign and date an informed consent form authorized by the relevant authorities.
5. The participation of the subject in another interventional study not interfering with the pathophysiological, pharmacological and clinical rationale of this protocol is possible.

Exclusion Criteria:

1. blood leukocytes >25 G/L.
2. Subject has already received anticancer treatment (drugs, surgery, radiotherapy) for AML, hematological malignancy or malignant cancer (within the last 2 years).
3. Subjects with AML with central nervous system involvement or promyelocytic type (AML-M3).
4. Subject to an uncontrolled intercurrent disease such as:

   * infection (viral, bacterial or fungal) requiring treatment;
   * symptomatic congestive heart failure;
   * unstable angina pectoris
   * cardiac arrhythmia
   * psychiatric illness or drug addiction that would limit compliance with study requirements (risk of treatment non-adherence or low venous capital).
5. Documented hypersensitivity to the drugs used to treat the subject.
6. Subject has been exposed to potent CYP450 inducers or inhibitors (including grapefruit, Seville oranges) within 7 days prior to treatment initiation.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with untreated AML and ineligible for standard cytarabine and anthracycline induction therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of mean plasma residual concentration of venetoclax | 1 month
  To compare the mean plasma residual concentration (ng/mL) of venetoclax (determined by LC-MS-MS) between patients who have entered composite complete remission (defined by the presence of remission criteria ≥ CRi, according to ELN 2022 guidelines) versus those who have not at the end of the first cycle of venetoclax+azacitidine treatment.

SECONDARY OUTCOMES:
Study relationship between mean plasma residual concentration of venetoclax and remission occurrence | 24 months
  To estimate mean residual plasma concentrations (Cres, ng/mL) of venetoclax and azole antifungals during patients' usual care. Then study the relationship between mean venetoclax Cres and the achievement (or non-achievement) of remission over time (according to ELN 2022 guidelines) .
Study performance of mean venetoclax Cres | 6 and 12 months
  To evaluate the performance (ROC curve) of mean venetoclax Cres (ng/mL) as a predictive biomarker of event-free survival (EFS) at 6 and 12 months.
Study survival | 24 months
  To estimate event-free survival (EFS), relapse-free survival (RFS) and overall survival (OS).
Study early deaths | 24 months
  To estimate the proportion of early deaths at 30 and 60 days post-inclusion.
Study the variability of plasma venetoclax and antifungal concentrations over time | 24 months
  To estimate the inter-individual (IIV) and intra-individual (IOV) variability of plasma venetoclax and antifungal concentrations over time.
Study the impact of parameters in uni- and multivariate analyses. | 24 months
  To estimate the impact of the following parameters to the diagnosis of remission or Cres (venetoclax):
  * patient characteristics: age [years], BMI ([kg/m²], sex[male vs female], ECOG [1,2 or 3], comorbidities reported in inclusion criteria, number of cytopenia grade>2, according to CTCAE v5, white blood cell count [G/L], creatininemia [µmol/L], cytoreduction (yes or not).
  * disease: AML classification (ELN 2022 guidelines), blast counts (G/L), cytogenetic status (fail, normal or not) and report, genetic status and report, abnormal rearrangement of genetic material and report.
  * and (co-)treatments of interest: fluconazole, isavuconazole, itraconazole, posaconazole, voriconazole, cannabidiol, ciclosporine, clarithromycine, diltiazem, ritonavir, verapamil,milk thistle, licorice; bosentan, carbamazépine, efavirenz, enzalutamide, felbamate, phénytoïne, phénobarbital, rifampicine, St. John's wort, grapefruit, bitter orange, star fruit).
Study adverse events of interest | 24 months
  To compare mean venetoclax Cres between patients who have experienced one or more of the 5 AEs of interest versus those who have not over time.

OTHER OUTCOMES:
ancillary study 1: study a medical device (VAMS Mitra, Neoteryx) to collect blood capillary sample as an alternative to venous puncture | 24 months
  To compare venetoclax Cres (ng/mL) values obtained with the Mitra® (Neoteryx) medical device (CE) with those obtained after conventional venipuncture (ng/mL).
ancillary study 2: study exposure of plasma venetoclax over 24h | 24 months
  To compute the total integrated area under the plasma venetoclax concentration-time curve (AUC) over 24h in 30 patients cared in CHU of Caen only and to identify the best time of sampling.
  Pharmacokinetic sampling (day 2 or 3 of cycle 2): Cres (prédose, ng/mL) and post-dose: 2h, 4h, 6h, 8h, 12h, 18h, 24h.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Marie Morice, PharmD, PhD, Principal Investigator — University Teaching Hospital of Caen; Sylvain Chantepie, MD, Principal Investigator — University Teaching Hospital of Caen
Locations (1):
- CHU de Caen, Caen, France